CLINICAL TRIAL: NCT06370117
Title: The Effects of Three Different Nonpharmacological Methods Used During Vascular Access in Children on Pain and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Bircan Kahraman Berberoglu, research asistant, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Aydın Adnan Menderes
Record Dates: First submitted 2024-04-04; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pain; Anxiety; Nurse's Role
Keywords: Pain; Anxiety; Nurse's Role; Child
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled experimental study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (n= 34) (No Intervention): Control group (n=34) Routine vascular access was performed on the children in the control group. Apart from this, no other application was made.
  Before the procedure; Introductory Information Form, Wong-Baker Facial Expression Rating Scale and Child Fear and Anxiety Scale were filled out by the researcher.
  Process order; Routine vascular access was performed. A stopwatch was used for the procedure time and the procedure time was recorded. The Child Fear and Anxiety Scale and the Wong-Baker Facial Expression Rating Scale were completed again.
- Buzzy Group (n= 34) (Experimental): Before the procedure; 60 seconds before starting the vascular access process, the Buzzy® tool was placed in the procedure area and cold and vibration application was started. The tourniquet was tied 10-12 cm above the vein to be treated. The Buzzy® tool was fixed to the middle part of the procedure area and the tourniquet, approximately 2 cm above the IV catheter entry site. As soon as the vascular access was established, the Introductory Information Form, Wong-Baker Facial Expression Rating Scale, and Child Fear and Anxiety Scale were filled out by the researcher. Process order; Application with the Buzzy® tool continued throughout the process. A stopwatch was used to time the procedure and the Buzzy® tool was removed when the procedure was completed. The Child Fear and Anxiety Scale and the Wong-Baker Facial Expression Rating Scale were completed again.
  Interventions: Behavioral: Buzzy
- Music video listening group (n= 34) (Experimental): The children in study group II were listened to music starting from 60 seconds before the vascular access procedure until the procedure ended.
  Before the procedure; A music video was played 60 seconds before starting the intravenous access procedure. The Introductory Information Form, Wong-Baker Facial Expression Rating Scale, and Child Fear and Anxiety Scale were filled in by the researcher.
  Process order; Music video playback continued. A stopwatch was used for the procedure time. As soon as the vascular access was established, the Child Fear and Anxiety Scale and the Wong-Baker Facial Expression Rating Scale were filled out again.
  Interventions: Behavioral: Music video listening
- Buzzy+ Music video listening Group (n= 34) (Experimental): Before the procedure; 60 seconds before starting the vascular access process, a music video was played and cold and vibration application was started with the Buzzy® tool.60 seconds before the procedure began, the Buzzy® tool was placed on the procedure area and cold and vibration application was initiated.Moreover,a music video was played. The tourniquet was tied 10-12 cm above the vein to be treated.The Buzzy® tool was fixed to the middle part of the procedure area and the tourniquet, approximately 2 cm above the IV catheter entry site. Introductory Information Form, Wong-Baker Facial Expression Rating Scale and Child Fear and Anxiety Scale were filled in by the researcher.Process order; application continued. A stopwatch was used for the procedure time.When vascular access was established, the Child Fear and Anxiety and Wong-Baker Facial Expression Rating Scale were filled out again.Once the process was finished, the buzzy was removed and the music video was closed.
  Interventions: Behavioral: Buzzy+ Music video listening

INTERVENTIONS:
Behavioral: Buzzy — Before the procedure; 60 seconds before starting the vascular access process, the Buzzy® tool was placed in the procedure area and cold and vibration application was started. The tourniquet was tied 10-12 cm above the vein to be treated. The Buzzy® tool was fixed to the middle part of the procedure area and the tourniquet, approximately 2 cm above the IV catheter entry site.
  Arms: Buzzy Group (n= 34)
Behavioral: Music video listening — Before the procedure; A music video was played 60 seconds before starting the intravenous access procedure.
  Arms: Music video listening group (n= 34)
Behavioral: Buzzy+ Music video listening — 60 seconds before starting the vascular access process, a music video was played and cold and vibration application was started with the Buzzy® tool. 60 seconds before the procedure began, the Buzzy® tool was placed on the procedure area and cold and vibration application was initiated. The tourniquet was tied 10-12 cm above the vein to be treated. The Buzzy® tool was fixed midway between the procedure area and the tourniquet, approximately 2 cm above the IV catheter entry site.
  Arms: Buzzy+ Music video listening Group (n= 34)

SUMMARY:
The research was conducted to evaluate the effects of three different non-pharmacological methods (playing a music video, buzzy application, listening to a music video + buzzy application) on the pain and anxiety levels of children in the 4-12 age group during vascular access.

H0.1. Playing music (music video) during the vascular access procedure has no effect on children's pain and anxiety levels.

H0.2. Applying buzzy during the vascular access procedure has no effect on children's pain and anxiety levels.

H0.3. Listening to a music video + applying buzzy during the vascular access procedure has no effect on children's pain and anxiety levels.

DETAILED DESCRIPTION:
Design: It is a randomized controlled experimental study. Methods: This study was conducted between February and December 2023 with 126 children between the ages of 4 and 12 who were hospitalized in the pediatric ward of a public hospital in a province in eastern Turkey and had vascular access. The sample consisted of four groups: a music video listening group (n=31), a buzzy group (n=32), a music video listening + buzzy group (n=31), and a control group (n= 32). Children were selected into groups by simple randomization method. Data were collected 60 seconds before starting the vascular access procedure and as soon as the procedure was completed. Introductory Information Form, Child Fear and Anxiety Scale and Wong-Baker Facial Expression Rating Scale were used to collect data.

The data was analyzed on SPSS (Version 25, Chicago, IL, USA). The Gaussian curve and Shapiro-Wilk test were used to assess whether or not the data were normally distributed. Descriptive statistical tests (arithmetic mean, standard deviation, number, and percentage) were also conducted. The conformity of the measurement values to normal distribution was tested with "Shapirow-wilk" analysis. Pearson chi-square test was applied to the dependency relationship of frequency measurement values. One-factor ANOVA test was used to compare whether there was a statistically significant difference between the means of independent groups. Kruskal Wallis H-Test was used to compare groups that did not show normal distribution. Mann Whitney U test was used in further analysis to determine the difference between two independent groups. Wilcoxon test was used to test the significance of the difference between the scores of two related measurements. P values <0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 4-12
* being willing to participate in the study,
* being accompanied by their parents (mother or father).

Exclusion Criteria:

* Failure to establish vascular access on the first try

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Facial Expression Rating Scale | From date of randomization (February 1, 2023) until the date of (December 30, 2023)/ for 9 months
  Wong-Baker Facial Expression Rating Scale (WB-FRS): It was developed by Wong and Baker in 1981. This scale is used to diagnose pain in children aged 3-18. This scale has six faces representing pain intensity, increasing from zero to five from left to right (0 points = very happy/no pain, 5 points = the most severe pain). The face on the far left has a smiling expression, indicating a pain-free state, while the face on the far right has a crying expression, corresponding to the most severe pain. The child is told to choose the face that best expresses his/her feelings.

SECONDARY OUTCOMES:
Children's Fear and Anxiety Scale | From date of randomization (February 1, 2023) until the date of (December 30, 2023)/ for 9 months
  Children's Fear and Anxiety Scale (CCAS): McMurtry et al. It was developed by in 2011. In this scale, the child is shown a picture containing five facial expressions rated between 0 and 4 points. While 0 indicates no fear and anxiety; 4 represents the highest fear and anxiety [0: neutral expression (no anxiety), 1: very little fear (very little anxiety), 2: some fear (some anxiety), 3: more fear (more anxiety), 4: possible shows the highest fear (severe anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: BIRCAN KAHRAMAN BERBEROĞLU, Study Chair — Aydın Adnan Menderes Univercity
Locations (1):
- Bircan Kahraman Berberoğlu, Aydin, AYDIN-efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No